CLINICAL TRIAL: NCT03058003
Title: Correlation Between Central Sensitization Inventory and Posturographic Data
Status: Completed | Type: Observational
Sponsor: Caps Research Network (Other)
Responsible Party: Sponsor
Other Study IDs: CI-IRB-20170124001
Record Dates: First submitted 2017-02-16; First posted 2017-02-20 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Central Nervous System Sensitization
Keywords: balance, postural; postural equilibrium; chronic pain; Chronic nonspecific low back pain; Fibromyalgia; Cervicogenic headache; Chronic tension type headache; Irritable bowel syndrome; Whiplash associated disorder; Temporomandibular disorder
MeSH Terms: conditions — Chronic Pain; Fibromyalgia; Post-Traumatic Headache; Irritable Bowel Syndrome; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: subjects suffering from chronic pain undergoing Posturography Evaluation and Central Sensitization Inventory
  Interventions: Diagnostic Test: Posturography Evaluation; Other: Central Sensitization Inventory
- Healthy: subjects self assessed to be in good health undergoing Posturography Evaluation and Central Sensitization Inventory
  Interventions: Diagnostic Test: Posturography Evaluation; Other: Central Sensitization Inventory

INTERVENTIONS:
Diagnostic Test: Posturography Evaluation — Posturography testing using the extended modified Clinical Testing of Sensory Integration in Balance (ext_mCTSIB) protocol: the subjects will be required to stand on a hard or compliant surface in a comfortable posture, feet shoulder width, with eyes open or closed, arms to the side and free to move, gazing forward, and breathing normally, with head straight, turned right or left, flexed or extended
  Other Names: Balance Testing; CAPS® Testing
Other: Central Sensitization Inventory — Standard chronic pain questionnaire: the subjects will be required to score each of the 25 items on a scale from 0 (never) to 4 (always)

SUMMARY:
To investigate the use of balance as a screening tool for Central Sensitization, a condition of the nervous system that is associated with the development and maintenance of chronic pain. This is done by comparing the scores of a gold standard screening tool (the Central Sensitization Inventory) with balance data.

DETAILED DESCRIPTION:
First, subjects will be asked to answer a brief medical questionnaire pertaining their general health status: since some of the subjects will be self-assessed to be "healthy" (no medical examination will be conducted to determine if this is indeed the case), the questionnaire will be used to determine if there are any possible known causes of poor balance performance. The questionnaire will not constitute an inclusion/exclusion criterion, it just has a classification purpose.

Subjects will then be asked to fill in the Central Sensitization Inventory (CSI), scoring each of the 25 items on a scale from 0 (never) to 4 (always).

Then, subjects will stand for 2 minutes on a compliant surface (a 4" tall foam cushion of known mechanical properties) to "learn" how to stand on it. Afterward, they will undergo posturography testing using the extended modified Clinical Testing of Sensory Integration in Balance (ext_mCTSIB) protocol: the subjects will be required to stand on a hard or compliant surface in a comfortable posture, feet shoulder width, with eyes open or closed, arms to the side and free to move, gazing forward, and breathing normally, with head straight, turned right or left, flexed or extended.

ELIGIBILITY:
Inclusion Criteria:

* Adults, self assessed to be in good health, or medically diagnosed with any of the following pathologies: Chronic nonspecific low back pain (CNSLBP), Fibromyalgia (FM), Cervicogenic Headche (CH), Chronic Tension Type Headache (CTT), Irritable Bowel Syndrome (IBS), Whiplash Associated Disorder (WAD), Temporomandibular Disorder (TMD)

Exclusion Criteria:

* Pregnant women will be excluded, as will be minors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults, self assess to be in good health or diagnosed with Central Nervous System Sensitization
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Stability Score | immediately after data collection
  The Stability Score (calculated as percentage ratio of the actual sway and the theoretical limit of stability) will be used to investigate if there is any difference between healthy controls and subjects affected by chronic pain. Statistical tools such t-tests and correlation coefficients will be used for assess if there is a difference between the two groups
CSI | immediately after data collection
  The sum of all the answers to the Central Sensitization Inventory will be used to investigate if there is any difference between healthy controls and subjects affected by chronic pain. Statistical tools such t-tests and correlation coefficients will be used for assess if there is a difference between the two groups

SECONDARY OUTCOMES:
CSI-SS | immediately after data collection
  Correlation between the Stability Score and the CSI result for each individual to determine if balance is an indicator of Central Nervous System Sensitization

CONTACTS AND LOCATIONS:
Overall Officials: Paul Noone, PhD, Principal Investigator — Caps Research Network
Locations (2):
- Innova Brain Rehabilitation, Marietta, Georgia, United States
- Small Street Clinic, Hampton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No